CLINICAL TRIAL: NCT05626933
Title: Anatomical Restoration Cleft Palate Technique (ARC) for Secondary Velopharyngeal Incompetence Post Cleft Palate Repair
Brief Title: Buccinator Myomucosal Flap With Furlow Palatoplasty and VPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, principal investigator, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 2222
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Velopharyngeal Insufficiency
MeSH Terms: conditions — Velopharyngeal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Buccinator myomucosal flap with Furlow palatoplasty (Experimental)
  Interventions: Procedure: Buccinator myomucosal flap with Furlow palatoplasty

INTERVENTIONS:
Procedure: Buccinator myomucosal flap with Furlow palatoplasty — Anatomical restoration concept using Buccinator myomucosal flap with Furlow palatoplasty is an effective technique for lengthening the palate and improving speech outcomes

SUMMARY:
Nasopharyngoscopic examination of the 20 patients with secondary VPI following 2 flap palatoplasty will be done for visualization of the velopharyngeal port, allowing assessment of the pattern and grade of velopharyngeal closure during speech and the presence or absence of a velopharyngeal gap and after VPI repair by Buccinator myomucosal flap with Furlow palatoplasty

ELIGIBILITY:
Inclusion Criteria:

* 5-6 years old children with previous treated complete cleft palate with 2 flap palatoplasty technique, nonsyndromic.
* lip and palate repair performed by one craniofacial surgeon

Exclusion Criteria:

* Patients with syndromic cleft lip.
* Bilateral cleft lip
* Patient older younger 5 years.
* Associated Cardiac anomalies.
* Any systemic condition

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-02 (Estimated)

PRIMARY OUTCOMES:
grade of velopharyngeal closure during speech | immediate postoperative
  Nasopharyngoscopic examination of the patients with secondary velopharyngeal insufficiency ( VPI) following two flap palatoplasty cleft palate repairs will be done for assessment of velopharyngeal closure grade during speech after VPI repair by Buccinator myomucosal flap with Furlow palatoplasty

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aboulhassan MA, Elrouby IM, Refahee SM, Abd-El-Ghafour M. Effectiveness of secondary furlow palatoplasty with buccal myomucosal flap in correction of velopharyngeal insufficiency in patients with cleft palate. Clin Oral Investig. 2024 Apr 17;28(5):257. doi: 10.1007/s00784-024-05607-4. PMID 38630186